CLINICAL TRIAL: NCT04660747
Title: Direct Oral Anticoagulants for the Treatment of Cerebral Venous Thrombosis: An International Phase IV Study
Brief Title: Direct Oral Anticoagulants for the Treatment of Cerebral Venous Thrombosis
Acronym: DOAC-CVT
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: University of Lisbon (Other); Sahlgrenska University Hospital (Other); University of Helsinki (Other); Centro Hospitalar de Lisboa Central (Other)
Responsible Party: Principal Investigator, Jonathan Coutinho, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: DOAC-CVT
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Venous Thrombosis
Keywords: Cerebral Venous Thrombosis; Cerebral Venous Sinus Thrombosis; Oral Anticoagulants; Direct Oral Anticoagulants; Vitamin K Antagonists
MeSH Terms: conditions — Intracranial Thrombosis | interventions — Anticoagulants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CVT cohort
  Interventions: Drug: Oral anticoagulant

INTERVENTIONS:
Drug: Oral anticoagulant — Direct oral anticoagulants or vitamin K antagonists. Please note that the study is fully observational. The choice of anticoagulant type and duration of treatment are left at the discretion of the treating physicians and patients. No treatment, intervention, or examinations are imposed on patients in the context of this study.

SUMMARY:
Rationale: Patients with cerebral venous thrombosis (CVT) are currently treated with anticoagulants during 3-12 months after diagnosis, to prevent worsening of the CVT and recurrent thrombosis, and to promote venous recanalization. Until recently, patients were generally treated with vitamin K antagonists (VKA). Direct oral anticoagulants (DOACs) are more practical in use than VKA and carry a lower risk of intracranial hemorrhage (ICH) in other conditions. One of the burning clinical questions is whether CVT patients can be safely treated with DOACs instead of VKA. In 2019, the first randomized trial on the safety and efficacy of DOACs in CVT was published (RESPECT-CVT). This exploratory study included 120 patients and the results suggest that DOACs can be safely used to treat CVT. Following RESPECT-CVT, use of DOACs to treat CVT is expected to rise, but given the limited sample size and strict selection criteria of RESPECT-CVT, additional data regarding the efficacy and safety of DOACs in CVT are required, especially from routine clinical care.

Objective: To assess the safety and efficacy of DOACs for the treatment of CVT in a real-world setting.

Study design: DOAC-CVT is an international, prospective, comparative cohort study. Initially, DOAC-CVT was designed to recruit 500 patients in a three-year study period. All patients recruited until January 15, 2024 will be included in the primary data analysis as previously described (https://doi.org/10.3389/fneur.2023.1251581). In addition, we will continue patient recruitment in an extension of the study until January 2026 to have a larger sample size, add new research questions, and to further strengthen global. We aim to recruit 1300 patients and anticipating a 3:2 ratio in DOAC:VKA use, we expect that in total 780 patients treated with a DOAC will be included.

Study population: Patients are eligible if they are >18 years old, have a radiologically confirmed CVT, have started oral anticoagulant treatment (DOAC or VKA) within 30 days of CVT diagnosis, and are included in the study within 90 days after CVT diagnosis.

Primary study endpoint: The primary endpoint is a composite of major bleeding (according to the criteria of the International Society on Thrombosis and Haemostasis) AND symptomatic recurrent venous thrombosis after 6 months of follow-up.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: This is an observational study which poses no risk or burden to the participant. Only data that are collected as part of routine clinical care will be used.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for the use of observational data
* Age >18 years at the time of CVT diagnosis
* Radiologically confirmed CVT diagnosis (CT-venography, MRI or catheter angiography)
* Oral anticoagulant treatment (DOAC or VKA) started within 30 days of CVT diagnosis (patient may initially be treated with heparin)
* Inclusion in the study within 90 days of CVT diagnosis

Exclusion Criteria:

* Anticoagulant treatment at the time of CVT diagnosis
* Pregnancy or lactation (post-partum women are eligible if they do not give breast-feeding)
* Mechanical heart valve
* Severe renal insufficiency (defined as an eGFR <15 ml/min)
* Severe liver disease resulting in clinically relevant coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with CVT treated at the participating centres. Both patients who are admitted to the hospital and patients who are treated via outpatient clinic are eligible. Centers participating in the DOAC-CVT study keep a log of all patients with CVT presented at their hospital during the study period to register which patients were included in the study and which patients were not eligible for inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Composite Outcome: Number of Participants with Major Bleeding and Recurrent VTE | Within 6 months after CVT diagnosis
  Major bleeding is defined according to the criteria of the International Society on Thrombosis and Haemostasis. Recurrent VTE is defined as symptomatic recurrent venous thromboembolism

SECONDARY OUTCOMES:
Mortality Rate | Within 3, 6, and 12 months after CVT diagnosis
  All-cause mortality
Number of Participants with Recurrent VTE | Within 3, 6, and 12 months after CVT diagnosis
  Symptomatic recurrent venous thromboembolism
Number of Participants with Major Bleeding | Within 3, 6, and 12 months after CVT diagnosis
  According to the criteria of the International Society on Thrombosis and Haemostasis
Number of Participants with Clinically Relevant Non-Major Bleeding | Within 3, 6, and 12 months after CVT diagnosis
  According to the criteria of the International Society on Thrombosis and Haemostasis
Number of Participants with Arterial Thrombotic Event | Within 3, 6, and 12 months after CVT diagnosis
Modified Rankin Scale | At 3, 6, and 12 months after CVT diagnosis
  Scale ranges from 0 to 6, with higher scores indicating worse functional outcome
Cerebral Venous Recanalization Rate | At 6 months after CVT diagnosis
  According to predefined criteria (see study protocol)
Frequency of chronic post-CVT symptoms | At 12 months after CVT diagnosis
  Outcome added in the extension study
Symptomatic recurrent VTE rate | At 24 months after CVT diagnosis
  Outcome added in the extension study

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Coutinho, MD, PhD, Principal Investigator — Amsterdam UMC, location AMC
Locations (1):
- Jonathan Coutinho, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van de Munckhof A, van Kammen MS, Tatlisumak T, Krzywicka K, Aaron S, Antochi F, Arauz A, Barboza MA, Conforto AB, Contreras DG, Heldner MR, Hernandez-Perez M, Hiltunen S, Ji X, Kam W, Kleinig TJ, Kristoffersen ES, Leker RR, Lemmens R, Poli S, Wasay M, Wu T, Yesilot N, Chen J, Cotelli MS, Demeestere J, Duan J, Ergin N, Freitas TE, Gomes A, den Hertog HM, Lindgren E, Martinez-Majander N, Metanis I, Miraclin A, Rani LJ, Reddy YM, Saleem S, Scutelnic A, Shanmugasundaram S, van den Wijngaard IR, Gencdal IY, van Eekelen R, Vellema J, Arnold M, Neto L, Middeldorp S, de Sousa DA, Jood K, Putaala J, Ferro JM, Coutinho JM; DOAC-CVT investigators. Direct oral anticoagulants versus vitamin K antagonists for cerebral venous thrombosis (DOAC-CVT): an international, prospective, observational cohort study. Lancet Neurol. 2025 Mar;24(3):199-207. doi: 10.1016/S1474-4422(24)00519-2. PMID 39986309
- [Derived] van de Munckhof A, Sanchez van Kammen M, Krzywicka K, Aaron S, Aguiar de Sousa D, Antochi F, Arauz A, Barboza MA, Conforto AB, Dentali F, Galdames Contreras D, Ji X, Jood K, Heldner MR, Hernandez-Perez M, Kam W, Kleinig TJ, Kristoffersen ES, Leker RR, Lemmens R, Poli S, Yesilot N, Wasay M, Wu TY, Arnold M, Lucas-Neto L, Middeldorp S, Putaala J, Tatlisumak T, Ferro JM, Coutinho JM. Direct oral anticoagulants for the treatment of cerebral venous thrombosis - a protocol of an international phase IV study. Front Neurol. 2023 Sep 14;14:1251581. doi: 10.3389/fneur.2023.1251581. eCollection 2023. PMID 37780701

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/47/NCT04660747/Prot_SAP_000.pdf